CLINICAL TRIAL: NCT04496674
Title: PPhase-I Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of the Bispecific PSMAxCD3 Antibody CC-1 as Single Agent and Combined With Checkpoint Blockade in Patients With Squamous Cell Carcinoma of the Lung
Brief Title: Bispecific PSMAxCD3 Antibody CC-1 in Patients With Squamous Cell Carcinoma of the Lung
Acronym: 2019-004849-32
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: premature termination of the trial due to bad recruitment
Sponsor: German Cancer Research Center (Other)
Collaborators: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-004849-32
Record Dates: First submitted 2020-05-08; First posted 2020-08-03 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancer Squamous Cell
Keywords: third line therapy; SCC; Metastatic squamous cell cancer
MeSH Terms: conditions — Neoplasms, Squamous Cell

STUDY DESIGN:
Intervention Model Description: Open-label, multicenter dose escalation and dose expansion phase I trial, designed to gain evidence of maximally tolerated and recommended phase-II dose of CC-1 in adult patients with SCC of the lung
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with bispecific Ab CC-1 (Experimental): administration of bispecific PSAMxCD3 Ab CC-1.
  Interventions: Drug: CC-1 and Toczilizumab

INTERVENTIONS:
Drug: CC-1 and Toczilizumab — Adminsitration of CC-1 and Toczilizumab

SUMMARY:
This trial is a phase I study in patients with metastatic non-small-cell lung cancer (NSCLC) after failure of second line therapy aiming to evaluate safety and efficacy of CC-1, a bispecific antibody (bsAb) with PSMAxCD3 specificity developed within DKTK. CC-1 binds to human prostate-specific membrane antigen (PSMA) on tumor cells of squamous cell carcinoma of the lung (SCC) as well as to tumor vessels of SCC, thereby allowing for a dual mode of anti-cancer action. CC-1 was developed in a novel format which not only prolongs serum half-life but most importantly reduces off-target T cell activation with expected fewer side effects. Together with preemptive IL-6 receptor (IL-6R) blockade using tocilizumab, this allows for application of effective bsAb doses with expected high anticancer activity. The study comprises two phases: The first phase is a dose-escalation phase with concomitant prophylactic application of tocilizumab to evaluate the maximally tolerated dose (MTD) of CC-1. This is followed by a dose-expansion phase (also with prophylactic IL-6R blockade using tocilizumab). A translational research program comprising, among others, analysis of CC-1 half-life and the induced immune response as well as molecular profiling in liquid biopsies will serve to better define the mode of action of CC-1 and to identify biomarkers for further clinical development.

DETAILED DESCRIPTION:
SCC of the lung is an aggressive malignant disease with poor prognosis after failure of established therapies. Any drug employed after second-line treatment is associated with only limited clinical benefit. Therefore, there is a high medical need for new therapeutic approaches in this patient population. The clinical effects of immune checkpoint inhibitors in NSCLC have proven the potential of T-cell based immunotherapy in this entity. The rationale for the therapeutic use of CC-1 is based on its proposed mode of action as a bsAb being specifically designed to direct T cells via its CD3 binding part towards tumor target cells via its PSMA binding part. Furthermore, CC-1 also reacts with tumor vessels of NSCLC thereby allowing for a dual mode of anti-cancer action by also attacking tumor blood supply and allowing for improved influx of immune effector cells. Due to its unique ability to redirect T cells via CD3 for PSMA-expressing tumor cell lysis, CC-1 can elicit repeated target cell elimination by cytotoxic T cells and a polyclonal response of previously primed CD4+ and CD8+ T cells. Compared to other immunotherapeutics presently being approved or in development (bsAbs with alternative formats like the authorised bsAb blinatumomab or other antibodies or CAR T cells), CC-1 is expected to offer the following major advantages:

(i) Reduction of off-target T cell activation and thus reduction of side effects due to its optimized format (ii) The possibility to tightly steer anti-target activity via serum level-controlled antibody application which, in contrast to CAR T cells, allows for termination of activity if desired.

On the background of the poor prognosis of patients with SCC of the lung after second-line therapy, the bsAb CC-1 holds promise as a new treatment option of immunotherapy for these patients.

The planned study will include patients with SCC of the lung with detectable PSMA expression on tumor cells after second line treatment. PSMA expression is to be determined by central immunohistochemical assessment of fresh or kryopreserved tumor samples. Only patients with proven PSMA expression on tumor cells as defined by ≥10% positivity of tumor cells can be included. The requirement of ≥10% positivity of tumor cells for PSMA expression cells is in line with definitions of positivity for target antigen expression employed for other antibodies used in cancer treatment, for example the human epidermal receptor protein-2 (HER2)-specific antibodies trastuzumab and pertuzumab. Both antibodies are approved for the treatment of HER2-positive breast cancer, and HER2 positivity is given if ≥10% of tumor cells show staining for HER2 as assessed by immunohistochemistry .

PSMA-positivity is estimated for about 50% of screened patients with SCC of the lung.

Further as a translational research program the investigators implemented PSMA-PET CTs at different time points. PSMA positivity in PSMA-PET CT has been described on several tumor entities including tumors of the lung. In line, PSMA expression has been described on tumor cells and neovasculature of tumor in lung cancer, especially SCC of the lung. However, a correlation of PSMA-PET positive tumors with immunhistochemical PSMA evaluation has so far not been described.

The implementation of PSMA-PET as additional imaging to routine CT, will further improve treatment for patients with SCC of the lung as results of PSMA-PET may replace biopsy in future patients. A maximum of three PSMA-PET CTs may be performed.

Study rationale with regard to objectives and further development of CC-1

In nonclinical studies, in vitro and in vivo, proof of concept, preliminary PK and PK/PD effects as well as toxicology have been evaluated. However, due to differences between animal models and the human situation, some aspects have to be assessed and further characterised in humans. For example, the target mediated drug disposition (TMDD), an effect that largely influences the serum half-life of antibody molecules particularly at low concentrations, cannot be properly addressed in mice. Furthermore, non-human primates (NHP) and rodents have several limitations as predictive models for toxicity and immunogenicity evaluation of CC-1. The CD3 binding part of CC-1 does not cross-react with CD3 of macaques and thus it is not possible to evaluate in these NHPs dose limiting side effects. Likewise, although CC-1 is cross-reactive with macaque-PSMA, PSMA distribution in macaques significantly differs from that in humans. The same holds true for rodents.

Due to the high medical need for patients with SCC of the lung after second-line treatment, the planned phase I trial is designed to confirm and further explore the safety and tolerability of the PSMAxCD3 bsAb CC-1 in adult patients with SCC of the lung. The primary objective is incidence and severity of adverse events (AEs) under therapy with CC-1. Furthermore, the trial aims to expand experience on pharmacokinetics, pharmacodynamics and toxicology of CC-1 from nonclinical studies to the human situation in relation to the PK, expected efficacy and safety. A focus will be on the following specific aspects/parameters:

* Pharmacokinetics and pharmacodynamics of CC-1 in humans
* Immunogenicity of CC-1 in humans based on both absolute (number and percentage of subjects who develop human anti-human antibody (HAHA).
* Absolute changes from baseline in laboratory parameters
* Change in cytokines from baseline
* Assessment of response rate by RECIST on routine imaging
* Evaluation of PSMA PET CT in a translational research program
* Overall and progression free survival

Rationale for preemptive IL-6R blockade by Tocilizumab

As described above, in the planned study the investigators exploit the strategy to use tocilizumab rather to prevent development of CRS in the first place than to treat CRS once it has arisen.

This strategy holds promise to increase the safety of study patients and timely study conduct. By starting the study treatment with CC-1 directly with prophylactic tocilizumab, all study patients will benefit from the expected advantage of this combination with regard to safety and can be treated with sufficiently high doses of CC-1 to achieve dose levels high enough to hopefully result in efficacy effects.

The rationale for preemptive IL-6R blockade by tocilizumab treatment is based on i. The firmly established efficiency and safety of tocilizumab for the treatment of CRS

ii. Lack of clear evidence for increased tumor growth as potential drawback of IL-6R blockage iii. Observations that IL-6 activity, while being responsible for the undesirable sequelae of CRS, appears not to be required for the therapeutic activity of CC-1 CRS that was induced by therapy with the approved bsAb blinatumomab was reported to be successfully treated by tocilizumab. Most importantly, despite rapid disappearance of clinical CRS symptoms, the therapeutic activity of the bsAb blinatumomab was maintained. Furthermore, tocilizumab was also used in the very recent FIH study with the REGN1917 (CD20xCD3) antibody.

Our own nonclinical studies demonstrate that tocilizumab does not impair the therapeutic activity of CC-1, neither in vitro nor in vivo. This is in contrast to steroids which are currently recommended and used as pre- and concomitant treatment to prevent CRS upon blinatumomab therapy.

Due to the mechanism of action of tocilizumab, there is a theoretical risk of tumor development or tumor progression due to immune modulation. On the basis of the current literature derived from large studies conducted in Japan, the USA and Europe, however, there is no evidence for an increased tumor risk upon application of tocilizumab. Only one Japanese study described a minimally increased risk of de novo lymphoma development. However, this could not be confirmed in any other study. Especially for lung cancer, there is no evidence for an increased incidence rate. Interestingly, high systemic IL-6 levels are associated with dismal prognosis in NSCLC. Furthermore, tocilizumab is currently being investigated in several Phase I/II studies for the treatment of solid and hematological neoplasia without evidence for an influence on tumor pathophysiology. Based on these findings, no relevant negative effects of tocilizumab on the efficacy and safety of CC-1 are expected.

ELIGIBILITY:
Inclusion Criteria:

* • Existence of a written informed consent

  * Patient is able to understand and comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations
  * SCC of the lung with detectable PSMA expression by tumor cells after second line treatment. PSMA expression is to be determined by central immunohistochemical assessment of fresh or cryopreserved tumor samples. Only patients with proven PSMA expression by tumor cells as defined by ≥10% positivity of tumor cells can be included.
  * Life expectance of > 3 months
  * At least one measurable lesion that can be accurately assessed at baseline by CT or MRI and is suitable for repeated assessment
  * Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2
  * Patient aged ≥ 18, no upper age limit
  * Female patients of child bearing potential and male patients with partners of child bearing potential, who are sexually active, must agree to the use of two effective forms (at least one highly effective method) of contraception. This should be started from the signing of the informed consent and continue throughout period of taking study treatment and for 1 month (female patients) / 3 months (male patients) after last dose of study drug. Postmenopausal or evidence of non-childbearing status. For women of childbearing potential: negative urine or serum pregnancy test within 21 days prior to study treatment and confirmed prior to treatment on day 1. Postmenopausal or evidence of non-childbearing status is defined as:
* Amenorrhoeic for 1 year or more following cessation of exogenous hormonal treatments
* Luteinizing hormone (LH) and Follicle stimulating hormone (FSH) levels in the post menopausal range for women under 50
* Radiation-induced oophorectomy with last menses >1 year ago
* Chemotherapy-induced menopause with >1 year interval since last menses
* Surgical sterilisation (bilateral oophorectomy or hysterectomy)

  * Adequate bone marrow, renal, and hepatic function defined by laboratory tests within 14 days prior to study treatment:

Neutrophil count ≥ 1,500/mm3 Platelet count ≥ 100,000/µl Bilirubin ≤ 1.5 x upper limit of normal (ULN) ALT and AST ≤ 2.5 x ULN PT-INR/PTT ≤ 1.5 x ULN Creatine kinase ≤ 2.5 x ULN Serum creatinine ≤ 1.5 mg/dl or creatinine clearance ≥ 60 ml/min

Exclusion Criteria:

* • Other malignancy within the last 5 years except: adequately treated non-melanoma skin cancer, carcinoma in situ of the cervix, carcinoma in situ of the breast, histological finding of prostate cancer of TNM stage T1

  * PSMA expression <10% by tumor cells
  * Concurrent or previous treatment within 30 days in another interventional clinical trial with an investigational anticancer therapy
  * Persistent toxicity (≥Grade 2 according to Common Terminology Criteria for Adverse Events [CTCAE] version 5.0) caused by previous cancer therapy, excluding alopecia and neurotoxicity (≤ 2 grade)
  * Clinical signs of active infection (> grade 2 according to CTCAE version 5.0)
  * Cerebral/Meningeal manifestation of the SCC of the lung
  * History of HIV infection
  * Immunocompromised patients
  * Viral active or chronic hepatitis (HBV or HCV)
  * History of autoimmune disease
  * History of relevant CNS pathology or current relevant CNS pathology (e.g. seizure, paresis, aphasia, cerebrovascular ischemia/hemorrhage, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, psychosis, coordination or movement disorder)
  * Epilepsy requiring pharmacologic treatment
  * Therapeutic anticoagulation therapy
  * Major surgery within 4 weeks of starting study treatment. Patients must have recovered from any effects of major surgery.
  * Patients receiving any systemic chemotherapy or radiotherapy within 2 weeks prior to study treatment or a longer period depending on the defined characteristics of the agents used
  * Heart failure NYHA III/IV
  * Severe obstructive or restrictive ventilation disorder
  * Known history of GI-perforation
  * Known intolerance to CC-1, tocilizumab or other immunoglobulin drug products as well as hypersensitivity to any of the excipients present in the respective drug products (CC-1, tocilizumab)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) (CTCAE V5.0) over 22 days | 10-72 patients. at least 1 cycle (for 22 day cycles) plus 21 days follow-up, but may vary depending on treatment-induced clinical benefit and optional additional cycles
  Incidence and severity of adverse events (AEs) (CTCAE V5.0) over 22 days (i.e. until end of first treatment cycle)
  Full hematology assessments for safety hemoglobin, red blood cells, platelets, mean cell volume, mean cell hemoglobin concentration, mean cell hemoglobin, white blood cells, absolute differential white cell count and absolute neutrophil count or segmented neutrophil count and Band forms should be performed at each visit and when clinically indicated.
  Biochemistry assessments for safety:
  sodium, potassium, calcium, magnesium, glucose, creatinine, total bilirubin, gamma glutamyltransferase, alkaline phosphatase,aspartate transaminase, alanine transaminase, urea or blood urea nitrogen, total protein, albumin and lactic dehydrogenase are performed.
Dose expansion part | 14 patients.at least 1 cycle (for 22 day cycles) plus 21 days follow-up, but may vary depending on treatment-induced clinical benefit and optional additional cycles
  To define the recommended phase-II dose of CC-1 under preemptive IL-6R blockade
  I

SECONDARY OUTCOMES:
Immunogenicity | day 15, day 43
  Number and percentage of subjects who develop HAHA at day 15 of every cycle and End Of Safety follw-up (day 43 of last cycle of a given patient) as compared to baseline.
  n case of CC-1 in this study, AESIs include cytokine-release syndrome (CRS) as the major "class toxicity" for bsAbs, anaphylactic reactions and immunogenicity of the drug substance
  With regard to trial schedule and AESI occurrence, AESIs constitute:
  * CRS (i.e. within treatment period)
  * Anaphylactic reactions upon study drug administration (i.e., within 24h)
  * Development of anti-CC-1 antibodies (HAHA) (day 15, day 43)
  AESIs are always be addressed as part of the patient safety report to the DSMB, also non-occurrence will be mentioned . Depending on severity of the AESI, dose reduction or discontinuation of treatment (DLT) may be necessary. Of note, allergic /anaphylactic reactions are not defined as DLT.
Anti-tumor activity | End of safety follow up,day 22 of cycle 3 and 4
  Objective tumor response assessed by RECIST on routine imaging at End of safety follow-up and thereafter for 12 months every 3 months.
  • For patients receiving more than one cycle objective tumor response will be assessed by RECIST on additional routine imaging every 6 weeks, i.e. prior to the application of cycle 3 (day 22 +/- 5 days of cycle 2) and cycle 5 (day 22 +/-5 days of cycle 4).
  Tumor response rate (TRR) The TRR is defined as the percentage of patients with complete remissions (CR) and partial remissions (PR) according to RECIST version 1.1. The TRR will be assessed at 3 and 6 months, as well as every 3 months during the extended treatment period (compare Trial Schedule). For patients receiving additional treatment cycles TRR will be assessed before the application of cycle 3 (day 22 +/- 5 days of cycle 2) and cycle 5 (day 22 +/-5 days of cycle 4).
Survival | 12 month after end of safety follow up
  OS is defined as the time from screening to time of death from any cause. Patients without event are censored at the last date of follow-up.

OTHER OUTCOMES:
PSMA PET CT | baseline, End Of safety follow up and at any timepoint dury study treatment if progressive disease is assumed in routine imaging
  Correlation with immunhistochemical proven PSMA expression on tumor at baseline
  • Value of PSMA-PET-CT in the context of treatment with CC-1 and progressive disease will be performed in terms of a translational research program to correlate PSMA expression as assessed by cryobiopsy with PSMA imaging. PSMA-PET CT will be performed at baseline, EOSf and at any time point during study treatment (cycle 1-6) if progressive disease is assumed in routine imaging, next imaging will be amended by PSMA-PET. Thus, a minimum of 2 and maximum of 3 PSMA-PET-CTs will be performed per patient.
Cytokine induction: | at baseline and at day 1-9, day 15 and day 22 in first cycle.
  Cytokines levels in serum as assessed
Pharmacokonteic | at day 1-9, day 15 and day 22 in the first cycle.
  CC-1 serum concentrations assessed

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Robert Bosch Centrum für Tumorerkrankungen, Stuttgart, Baden-Wurttemberg
  - University Hospital Tuebingen, CCU Translational Immunology, Tübingen, Baden-Wurttemberg